CLINICAL TRIAL: NCT06231459
Title: Expression of Pro- and Anti-inflammatory Cytokines During Anti-PCSK9 Therapy in Patients With Statin-resistant Familial Hypercholesterolemia
Brief Title: Expression of Pro- and Anti-inflammatory Cytokines During Anti-PCSK9 in Familial Hypercholesterolemia
Acronym: CytoEx-PCSK9
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Juan Antonio Suárez Cuenca, MD, PhD, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 061.2019
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-controlled, before-after comparison, quasiexperimental, single-center study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evolocumab (Experimental): Evolocumab 140 mg was administered intramuscularly every two weeks at the discretion of their physiciansm according to LDLc response.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Evolocumab 140 mg was administered intramuscularly every two weeks at the discretion of their physiciansm according to LDLc response. Clinical-demographic and anthropometry data were collected during a direct interview. Blood sample was processed to obtain glycated hemoglobin complete blood count and serum lipids. Likewise, flow cytometry was used to characterize baseline circulating M1-, M2-macrophages and monocytes. Multiplexing of plasma samples was used to compare plasma fraktaline, IL-1, IL-4, IL-6, IL-8, IL-10, MCP-1 and TNF-alpha. Endpoints consisted of: 1) lower serum lipids; 2) modification of pro-inflammatory mediators (neutrophils, lymphocytes, NtLR, soluble pro-inflammatory cytokines).
  Other Names: repatha

SUMMARY:
Statins have been shown to reduce LDL cholesterol (LCLc) levels, stabilizing atheromatous plaque, reversing endothelial dysfunction and decreasing thrombogenesis. Novel pharmacological approaches, such as PCSK9 inhibitors (PCSK9i), effectively reduce LDL-c. In the clinical setting, there are cases of dyslipidemia showing lack of response to statin, known as statin-resistant familial hypercholesterolemia (SR-FH), where patients maintain a high cardiovascular risk despite statin therapy. Then, therapeutic alternatives are required. PCSK9i has shown to reduce cholesterol levels and risk of cardiovascular disease, particularly in patients with statin-resistant familial hypercholesterolemia; and recently, it has been hypothesized that PCSK9i have an effect on inflammation. Aim. To evaluate the effect of anti-PCSK9 treatment on markers related to the inflammatory response in patients with SR-FH.

Methods. Non-randomized, non-controlled, before-after comparison, quasiexperimental, single-center study on patients older than 18 years, with diagnosis statin-resistant FH (SR-FH), who were attended at the Cardiology Department, Centro Médico Nacional "20 de Noviembre ISSSTE", Mexico City. SR-FH was defined as symptomatic cardiovascular disease accompanied by LDL-C concentration higher than 160 mg/dL despite maximally tolerated statin dose. Clinical-demographic and anthropometry data were collected during a direct interview. Blood sample was processed to obtain glycated hemoglobin complete blood count and serum lipids. Likewise, flow cytometry was used to characterize baseline circulating M1-, M2-macrophages and monocytes. Multiplexing of plasma samples was used to compare plasma fraktaline, IL-1, IL-4, IL-6, IL-8, IL-10, MCP-1 and TNF-alpha. Endpoints consisted of: 1) lower serum lipids; 2) modification of pro-inflammatory mediators (neutrophils, lymphocytes, NtLR, soluble pro-inflammatory cytokines). Quatitative data were resumed as mean ± SD; while categorical data as n(%).One-way T-test was applied. Statistical significance was considered if p <0.05.

DETAILED DESCRIPTION:
Study Design Non-randomized, non-controlled, before-after comparison, quasiexperimental, single-center study.

Study Population Patients older than 18 years, with diagnosis statin-resistant FH (SR-FH), who were attended at the Cardiology Department, Centro Médico Nacional "20 de Noviembre ISSSTE", Mexico City. SR-FH was defined as symptomatic cardiovascular disease accompanied by LDL-C concentration higher than 160 mg/dL despite maximally tolerated statin dose (Ito MK, McGowan MP, Moriarty PM. Management of familial hypercholesterolemias in adult patients: recommendations from the National Lipid Association Expert Panel on Familial Hypercholesterolemia. J Clin Lipidol. 2011;5(3 Suppl):S38-S45. doi: 10.1016/j.jacl.2011.04.001.). We excluded patients with infections, neoplasia or under oncological therapy. The study was approved by the Research, Biosafety and Ethics Committee of the Centro Médico Nacional 20 de Noviembre ID 061.2019.

Clinical-Demographic characteristics Clinical-demographic characteristics like age, gender, past diseases and medication use were collected from a direct interview and verified through the medical record. Body mass index (BMI) was calculated as weight/height2 (kg/m2). Blood pressure was obtained while the patient was in a seated position and was considered to be the mean of three readings taken 5 min apart using a Welch Allyn 767 mobile aneroid sphygmomanometer (Welch Allyn Inc.; Skaneateles Falls, NY, USA). Diabetes Mellitus was defined according to the guidelines from the American Diabetes Association with one of the following conditions (repeated for confirmation at a separate date): 1) Hb A1C ≥ 6.5%; 2) fasting glucose ≥ 126 mg/dl; or 3) 2-h plasma glucose ≥ 200 mg/dl during an oral glucose tolerance test.

Complete Blood Count and Lipid Profile Following a 12-h fast, venous blood samples (4 ml) were collected into BD Vacutainer® tubes (Becton, Dickinson & Co., Franklin Lakes, NJ, USA) containing 1.8 mg ethylenediaminetetra-acetic acid/ml of blood. Standard blood cell count was performed immediately. For clinical chemistry blood simple was centrifuged at 1 200 g for 5 min, at 4°C, separated into fractions and plasma was stored at -80°C prior to analyses. Blood cell count and plasma triglycerides, total cholesterol, high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C) were determined using routine clinical laboratory equipment and a standard auto-analyser (Synchron CX®9 PRO Clinical System; Beckman Coulter, Brea, CA, USA). Atherogenic index was calculated as log triglyceride / HDL-C.

Flow Cytometry Blood sample was processed following standardized protocol; then, centrifuged to obtain leucocyte population. After three washes, cells were fixed in 4% paraformaldehyde and stored for 12 hours. Flow cytometry analysis (MACSQuant Analyzer 10 - Miltenyi Biotec) was performed in a total of 1,000,000 events collected for each analysis, and corresponding isotype controls were used to set appropriate regions. Cells subpopulations were identified by their specific marker combination (CD14+, CD163+ for M1-macrophages; CD14+, CD206+ for M2-macrophages; CD16+, CXCR4 receptor and CD16+, CXCR2 for monocytes.

Plasma Soluble Biomarkers An aliquot of blood sample was immediately centrifuged at 5000rpm/5 min and plasma was collected. Analytes (fraktaline, IL-1, IL-4, IL-6, IL-8, IL-10, MCP-1 and TNF-alpha), using commercially available multiplexing assay (HCYTOMAG-60-08K, MILLIPLEX MAP Human Cytokine/Chemokine Magnetic Bead Panel - Immunology Multiplex Assay Merc, Millipore Massachusetts, USA), and following manufacturer instructions; and read in Multiplex reader (MAGPIX System, Millipore, Austin, Texas).

Follow up and Study Endpoints Follow-up was conducted after 6 months of therapy, through programmed medical evaluations and blood analyses. Primary endpoint consisted of modification in: 1) serum lipids; while secondary end points included: 1) pro-inflammatory mediators (neutrophils, lymphocytes, NtLR, soluble pro-inflammatory cytokines); and 2) atherogenic index.

Statistical analysis

Quatitative data were resumed as mean ± SD; while categorical data as n(%).One-way T-test was applied. Statistical significance was considered if p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, with diagnosis statin-resistant FH (SR-FH), who were attended at the Cardiology Department, Centro Médico Nacional "20 de Noviembre ISSSTE", Mexico City. SR-FH was defined as symptomatic cardiovascular disease accompanied by LDL-C concentration higher than 160 mg/dL despite maximally tolerated statin dose

Exclusion Criteria:

* We excluded patients with infections, neoplasia or under oncological therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Asked self-representation of gender identity.
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
lower of serum lipids | 1 month
  lower serum LDL below 100mg/dL

SECONDARY OUTCOMES:
modification of pro-inflammatory mediators | 1 month
  modification of pro-inflammatory mediators, like neutrophils, lymphocytes, NtLR, soluble pro-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Julieta D Morales-Portano, MD, Principal Investigator — Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Locations (1):
- National Medical Center "20 de Noviembre", ISSSTE, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Possible data share but require institutional permission.

REFERENCES:
- [Background] D'Onofrio N, Prattichizzo F, Marfella R, Sardu C, Martino E, Scisciola L, Marfella L, Grotta R, Frige C, Paolisso G, Ceriello A, Balestrieri ML. SIRT3 mediates the effects of PCSK9 inhibitors on inflammation, autophagy, and oxidative stress in endothelial cells. Theranostics. 2023 Jan 1;13(2):531-542. doi: 10.7150/thno.80289. eCollection 2023. PMID 36632236